CLINICAL TRIAL: NCT02962310
Title: An Open Label, Randomized, 2-Period, 2-Treatment,2-Sequence, Crossover, Single-Dose BE of Rosuvastatin Ca Tab 40 mg [Torrent,India] Versus Crestor 40 mg Tab [ AstraZeneca Pharmaceuticals LP, USA] in Healthy Subjects-Fasted Condition.
Brief Title: Bio Equivalence Study of Torrent Pharmaceutical Ltd's Rosuvastatin Calcium Tablets Under Fasting Condition.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK-09-045
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (Experimental): Torrent Pharmaceutical Ltd's Rosuvastatin Calcium Tablets 40 mg
  Interventions: Drug: Torrent's Rosuvastatin Calcium Tablets 40 mg
- Reference (Active Comparator): Crestor 40 mg Tablets of AstraZeneca Pharmaceuticals LP, USA
  Interventions: Drug: Crestor 40 mg Tablets of AstraZeneca LP, USA

INTERVENTIONS:
Drug: Torrent's Rosuvastatin Calcium Tablets 40 mg — oral, crossover
  Arms: Test
Drug: Crestor 40 mg Tablets of AstraZeneca LP, USA — oral, crossover
  Arms: Reference

SUMMARY:
Subjects to compare the single dose bioavailability of Torrent's Rosuvastatin Calcium Tablets 40 mg and Crestor® 40 mg Tablets of AstraZeneca Pharmaceuticals LP, USA. Dosing periods of studies were separated by a washout period of 7 days.

DETAILED DESCRIPTION:
An Open Label, Randomized, 2-period, 2- Treatment, 2-Sequence, Crossover, Single-dose Bioequivalence Study of Rosuvastatin Calcium Tablets containing Rosuvastatin Calcium 40 mg ( Test Formulation, Torrent Pharmaceutical Ltd., India) Versus Crestor® 40 mg Tablets containing Rosuvastatin Calcium 40 mg (Reference , AstraZeneca Pharmaceuticals LP, USA) in Healthy Human Volunteers Under Fasting Condition.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* Age: 18-45 years
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day.

Exclusion Criteria:

* The volunteers were excluded from the study based on the following criteria:
* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute. Oral temperature less than 95°P or more than 98.6°P.
* Respiratory rate less than 12/minute or more than 20/minute
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* History of alcohol or drug abuse
* Positive breath alcohol test
* Recent history of kidney or liver dysfunction.
* History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of heart failure.
* HIV, HCV, HBsAg positive volunteers.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, Cocaine positive volunteers based on urine test.
* Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
* Administration of any study drug in the period 0 to 3 months before entry to the study.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* History of pre-existing bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose to 96 hours post-dose
AUC | Pre-dose to 96 hours post-dose

IPD SHARING:
Plan to Share IPD: No